CLINICAL TRIAL: NCT05555264
Title: Enhancing Impact of Internet-delivered Cognitive Behaviour Therapy for Alcohol Misuse by Addressing Co-morbidity and Improving Patient Narratives: a Patient-Oriented Research Approach
Brief Title: Enhancing Internet-delivered Cognitive Behaviour Therapy for Alcohol Misuse
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-082
Record Dates: First submitted 2022-08-08; First posted 2022-09-26 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Misuse
Keywords: Internet-delivered cognitive behaviour therapy; Alcohol misuse; Substance misuse; Patient Narratives; Co-morbidities

STUDY DESIGN:
Intervention Model Description: Each client will choose one of the following: self-guided Alcohol Change Course Enhanced (8 weeks), therapist-guided Alcohol Change Course Enhanced (8 weeks)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Guided Alcohol Change Course Enhanced (Experimental): Clients who select or are assigned the self-guided condition will receive access to 6 ICBT core lessons, 6 associated worksheets to enhance skill acquisition, and 8 additional resources addressing potential co-morbid concerns (e.g., Addressing Anger, Improving Assertiveness and Communication, Changing Cannabis Use, Developing Cognitive Coping, Coping with Grief, Understanding PTSD, Improving Sleep Quality, and Managing Worry). The 6 lessons and 6 associated worksheets are released at a rate of 1 per week over 7 weeks, with no new content being released to participants in Week 4. The 8 additional resources are available at any time during the course.
  Clients will not receive therapist support/guidance during the 8-week intervention.
  Interventions: Behavioral: Self-Guided
- Therapist-Guided Alcohol Change Course Enhanced (Experimental): Clients who select the therapist-guided condition will receive access to 6 ICBT core lessons, 6 associated worksheets to enhance skill acquisition, and 8 additional resources addressing potential co-morbid concerns (e.g., sleep quality, cannabis use). The 6 lessons and 6 associated worksheets are released at a rate of 1 per week over 7 weeks, with no new content being released to participants in Week 4. The 8 additional resources are available at any time during the course.
  Clients will receive therapist support/guidance during the 8-week intervention.
  Interventions: Behavioral: Therapist-Guided

INTERVENTIONS:
Behavioral: Self-Guided — Clients who select or are assigned the self-guided condition will be able to contact the Online Therapy Unit regarding any technical issues through the secure treatment platform; monitoring staff will respond by secure message to messages received however, no psychological intervention will be provided by monitoring staff as part of the ACCE treatment intervention. If there is a significant clinical issue requiring attention (e.g., a sudden increase in symptoms) monitoring staff will make a telephone call and crisis support will be provided if necessary.
  Arms: Self-Guided Alcohol Change Course Enhanced
Behavioral: Therapist-Guided — Therapists will spend ~15 minutes/week communicating with each client who selects the therapist-guided condition, primarily using secure messages. Phone calls will only be made if there is a significant clinical issue requiring attention that the therapist does not feel can be addressed in a message (e.g., a question about the materials that cannot be easily addressed in a text format, a sudden increase in symptoms, increased suicide risk).
  Arms: Therapist-Guided Alcohol Change Course Enhanced

SUMMARY:
Alcohol misuse is a common and disabling problem and refers to alcohol consumption that causes harm to the drinker, others, and/or greater society.

Internet-delivered cognitive behaviour therapy (ICBT) shows considerable promise as a convenient treatment for alcohol misuse. The overall goal of ICBT for alcohol misuse is typically behavioural change, measured in terms of reduction of drinks consumed, as opposed to abstinence. These interventions can be delivered in a therapist-guided format or self-guided format.

In past research on ICBT for alcohol misuse, stakeholders (e.g., patients, providers, and academics) highlighted the importance of ensuring that ICBT meets the needs of diverse residents of Saskatchewan, and that ICBT takes into account factors such as psychological comorbidity. Therefore, the goals of the current trial are to: 1) incorporate additional patient narratives to assist clients in learning how diverse individuals apply skills to their lives; and 2) provide additional optional resources to address potential co-morbid concerns. The study aims to examine how these materials are evaluated by clients. Furthermore, we will also examine the overall engagement and outcomes of the enhanced ICBT course for alcohol misuse benchmarked with past findings.

DETAILED DESCRIPTION:
In Canada, it is estimated that 16.6% of individuals over the age of 12 engage in heavy drinking on a monthly basis. The cost of alcohol misuse is substantial, as it is associated with psychological distress, interpersonal problems, chronic health conditions, health care costs, and lost work productivity. Unfortunately, the under treatment of alcohol misuse is a significant problem, with many individuals with alcohol misuse never seeking treatment, for reasons such as stigma or lack of available services due to rural and/or remote location.

Internet-delivered cognitive behaviour therapy (ICBT) for alcohol misuse is a growing and impactful method of effectively delivering care that overcomes several barriers of face-to-face therapy. Reflecting this trend, ICBT for alcohol misuse has been funded by the Saskatchewan Ministry of Health since July 2019. Specifically, the government funds the Online Therapy Unit (OTU) to deliver the Alcohol Change Course (ACC) to SK residents. In addition to the ACC, the OTU has delivered ICBT treatment programs addressing anxiety, depression, and various health conditions to over 10418 clients since 2010.

While there is growing recognition of the effectiveness of ICBT, there is also awareness of the need to improve ICBT for alcohol misuse to increase the impact of this innovative treatment approach.

Research suggests that the integration of patient suggestions can improve the quality of care, by ensuring that programs are designed in such a way that they are acceptable to patients and fit with other services; when this approach is taken, there is evidence that services are more effective and more likely to be used and sustained longer-term. Through such a patient-oriented process employed by the OTU in their research and development of the ACC, two opportunities for improving the ACC were identified (i.e., 1 - refining the existing patient narratives and incorporating new patient narratives to be more diverse in nature; and 2 - providing optional additional resources to address common comorbid concerns).

1. Patient narratives (referred to as "Personal Reflections" in the ACCE) are incorporated in ICBT programs to motivate and support health-behaviour change. They are typically brief descriptions of an individual, challenges they face, and their strategy use. Research supports the efficacy of patient narratives for providing information, engaging clients in behavioural change, modeling behaviour, and comforting clients. To capture the diverse characteristics and experiences (e.g., alcohol use, age, location of residence, gender, ethnicity) of future ACCE clients, the ACC's personal reflections were revised, and new personal reflections were developed.
2. Given high comorbidity of alcohol misuse and various concerns (e.g., depression, anxiety, PTSD, cannabis use, relationship troubles, anger, etc.), both past ACC clients and OTU therapists indicate the benefits of broadening the topics covered by additional resources in the ACCE. As such, eight ACCE-specific additional resources were offered as part of the ACCE, including Addressing Anger, Improving Assertiveness and Communication, Changing Cannabis Use, Developing Cognitive Coping, Coping with Grief, Understanding PTSD, Improving Sleep Quality, and Managing Worry.

In this study, prospective clients may learn of the ACCE from providers/organizations, who will be informed through posters, emails, and phone calls. Clients interested in the ACCE will be directed to the study website to complete a consent form explaining the screening protocol. Once clients give consent, they will complete an online screening questionnaire assessing eligibility and capturing demographic, contact, alcohol use, and other information. After completing the screening, clients will book a telephone screening interview with unit staff through the online appointment booking software. During the telephone screening, clients will be asked follow-up questions to confirm their eligibility. (If clients meet the current trial's exclusion criteria, they will be referred to more appropriate mental health services in their area).

At the end of the telephone screening, Saskatchewan clients who meet eligibility criteria will indicate their preference for the therapist-guided or self-guided (with monitoring) ACCE; screening staff will enroll them in the chosen course. Clients from outside Saskatchewan will be offered self-guided ACCE only. All enrolled clients will receive a username and temporary password, and will be informed that they can access the ACCE on the following Monday.

Once clients log onto the treatment platform, they will complete a pre-treatment questionnaire and a consent form explaining the nature of treatment. All clients will receive the ACCE. Lesson content is based on cognitive behaviour therapy and relapse prevention. Materials are presented in a didactic and case-enhanced learning format.

Participants will complete online questionnaires at various times as outlined below. At mid-treatment and/or post-treatment, a subsample of clients will be invited for semi-structured interviews to discuss their experiences with the revised personal reflections and additional resources. A research associate will monitor client demographics to ensure that a diverse sample is represented in the interviews, and may directly reach out to clients with diverse demographic or clinical characteristics.

ELIGIBILITY:
Inclusion Criteria:

* are residing in Saskatchewan;
* are over the age of 17;
* endorse alcohol misuse;
* and have access to a computer and the Internet.

Exclusion Criteria:

* have a severe medical condition and/or psychiatric illness (e.g., psychosis);
* show signs of severe depression;
* are assessed as being at high risk of suicide;
* have severe problems with drugs (other than alcohol and/or cannabis; measured by scoring > 24 on the DUDIT, or by clinical assessment);
* have severe cognitive impairment;
* demonstrate low motivation or concerns regarding completing the online treatment program;
* or do/will engage in ongoing or impending significant mental health treatment (i.e., >2 visits per month).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Drinks Preceding Week as Measured by Timeline Followback (TLFB) | Baseline (screening), Week 4 (mid-treatment), Week 7 (post-treatment), Week 20 (follow-up)
  Change in preceding week alcohol consumption in terms of the total number of standard drinks consumed on each day during the previous 7 days.
Heavy Drinking Days Preceding Week as Measured by Timeline Followback (TLFB) | Baseline (screening), Week 4 (mid-treatment), Week 7 (post-treatment), Week 20 (follow-up)
  Change in preceding week alcohol consumption in terms of the total number of heavy drinking days during the previous 7 days.
Patient Reflections Questionnaire | Week 4 (mid-treatment), Week 7 (post-treatment)
  Change in clients' opinions of and satisfaction with the personal reflections incorporated throughout the ACCE. This questionnaire has been developed by the research team, and does not have a sum score.
Additional Resources Questionnaire (Midpoint) | Week 4 (mid-treatment)
  Clients' opinions of and satisfaction with the 8 additional resources offered alongside the ACCE that they have reviewed since the beginning of treatment. This questionnaire has been developed by the research team, and does not have a sum score.
Additional Resources Questionnaire | Week 8
  Clients' opinions of and satisfaction with the 8 additional resources offered alongside the ACCE that they have reviewed since the Midpoint questionnaire. This questionnaire has been developed by the research team, and does not have a sum score.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9-item (PHQ-9) | Baseline (screening), Week 1, Week 4 (mid-treatment), Week 7 (post-treatment), Week 20 (follow-up)
  Change in depression symptoms. 9 items are summed into a total score, ranging from 0-27. Higher scores indicate higher depression severity.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline (screening), Week 7 (post-treatment), Week 20 (follow-up)
  Change in anxiety symptoms. 7 items are summed into a total score, ranging from 0-21, with higher scores indicating more severe self-reported levels of anxiety.
Alcohol Use Disorder Identification Test (AUDIT) | Baseline (screening), Week 7 (post-treatment), Week 20 (follow-up)
  Change in alcohol-related problems and behaviours measured via a total AUDIT score, which can range from 0-40. Greater scores indicate greater alcohol problems.
Penn Alcohol Craving Scale | Baseline (screening), Week 7 (post-treatment), Week 20 (follow-up)
  Change in alcohol craving measured via a total score ranging between 0-30. Higher scores indicate greater alcohol craving.
The Cannabis Use Disorder Identification Test - Revised (CUDIT-R) | Baseline (screening), Week 7 (post-treatment), Week 20 (follow-up)
  Change in cannabis-related problems and behaviours measured via total CUDIT-R score, which can range from 0-32 (8 items). Scoring >7 indicates hazardous cannabis use; scoring >11 indicates a possible cannabis use disorder.
Couples Satisfaction Index 4-item (CSI-4) | Baseline (screening), Week 7 (post-treatment), Week 20 (follow-up)
  Change in relationship satisfaction. Higher total scores indicate greater relationship satisfaction, with scores <13.5 indicating notable dissatisfaction.
Dimensions of Anger Reactions (DAR-5) | Baseline (screening), Week 7 (post-treatment), Week 20 (follow-up)
  Change in self-reported anger problems. Higher total scores indicate greater severity of anger problems. Scores range from 0-20.
Credibility and Expectancy Questionnaire (CEQ) | Week 4 (mid-treatment)
  Measures treatment credibility via the first 3 items (ranging from 1-9) from the CEQ. Total scores range from 3-27, with higher scores indicating higher perceived treatment credibility.
Open-Ended Personal Reflections and Additional Resources Questionnaire | Week 4 (mid-treatment)
  Measures client's feedback regarding the ACCE's enhanced personal reflections and additional resources, via a structured interview process. The number of participants to be interviewed will be determined based on the saturation of themes yielded within preliminary qualitative analyses. The structured interview questions were created by the research team and the measure does not have a sum score.
Open-Ended Personal Reflections and Additional Resources Questionnaire | Week 7 (post-treatment)
  Measures client's feedback regarding the ACCE's enhanced personal reflections and additional resources, via a structured interview process. The number of participants to be interviewed will be determined based on the saturation of themes yielded within preliminary qualitative analyses. The structured interview questions were created by the research team and the measure does not have a sum score.
Change Goal Questionnaire | Week 2, Week 7 (post-treatment)
  Change in clients' goals related to their alcohol use. This brief questionnaire has been developed by the research team, and does not have a sum score.
(Treatment Satisfaction) Evaluation Questions and Negative Effects | Week 7 (post-treatment)
  Measures negative effects experienced by clients during treatment. This questionnaire has been developed by the research team, and does not have a sum score.
Other Forms of Help | Week 7 (post-treatment), Week 20 (follow-up)
  Change in other types of help that clients received during treatment. This questionnaire has been developed by the research team, and does not have a sum score.
Insomnia Severity Index (ISI) | Baseline (screening), Week 7 (post-treatment), Week 20 (follow-up)
  Change in insomnia severity. 7 items assess clients' difficulties falling asleep, staying asleep, and waking too early, each on a scale from 0 (None) to 4 (Very Severe). Total scores range from 0-28.
Life Events Checklist for Diagnostic and Statistical Manual of Mental Disorders-5/PTSD Checklist for DSM-5 (LEC-5/PCL-5) | Baseline (screening)
  Measures PTSD symptoms. The LEC-5 is a checklist of common traumatic events used to establish the nature of the traumatic events a client has experienced. This questionnaire is not intended to be scored, but is used for descriptive purposes. Following the LEC-5, clients will complete the PCL-5 (a validated measure of PTSD, based on DSM-5 criteria); PCL-5 scores range from 0-80, and higher total scores indicate greater PTSD severity.
Short Form PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders-5 (SF-PCL-5) | Week 7 (post-treatment), Week 20 (follow-up)
  Change in PTSD symptom severity. The SF-PCL-5 is A 4-item, short-form version of the PTSD Checklist for DSM-5. Higher total scores indicate greater PTSD severity. Scores range from 0-16.
Motivation for Change | Baseline (screening), Week 4 (mid-treatment), Week 7 (post-treatment)
  Change in clients' motivation for changing their alcohol use. On three scales from 1-10, clients self-report: 1) the importance of changing their alcohol use, 2) their confidence in their ability to change their alcohol use, and 3) their readiness to change their alcohol use.
Work and Social Adjustment Scale (WSAS) | Baseline (screening), Week 7 (post-treatment), Week 20 (follow-up)
  Change in impairment of functioning. Measure includes 5 questions assessing impairment of functioning. Items are scored on a scale of 0 to 8. Total scores on the WSAS range from 0 to 40 with higher scores suggesting severe impairment.
Total Drinks in the Last Week | Week 1, Week 2, Week 3, Week 5, Week 6, Week 8
  Description: Change in preceding week alcohol consumption in terms of the total number of standard drinks consumed on each day during the previous 7 days.

OTHER OUTCOMES:
Family History Density - Alcohol (FHD-Alcohol) | Baseline (screening)
  Measures clients' family history density of alcohol use and alcohol-related difficulties via 6 items. Total scores range from 0-2; higher scores indicate a greater family history density of alcohol use and alcohol use-related difficulties.
Drug Use Disorder Identification Test (DUDIT) | Baseline (screening)
  Measures problematic drug use via an 11-item screening tool. Items 1-9 are scored on a scale ranging from 0-4. Items 10 and 11 are scored as a 0, 2, or 4. Total scores for the DUDIT range from 0-44, with higher scores suggesting more problematic drug use.
Homework Reflection Questionnaire | Weeks 2-8
  Measures clients' week-to-week experience in the ACCE. This brief questionnaire has been developed by the research team, and does not have a sum score.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada